CLINICAL TRIAL: NCT02853227
Title: The Telemark Breast Score is a Valid Method for the Evaluation of Outcome After Reconstructive Surgery of the Breast
Brief Title: The Telemark Score: a Reliable Method for Evaluation of Results After Breast Surgery
Acronym: TBS
Status: Completed | Type: Observational
Sponsor: Sykehuset Telemark (Other Government)
Responsible Party: Principal Investigator, Anadi Begic, overlege, Sykehuset Telemark
Other Study IDs: 1097.13-1; 2013/1197 (Other: REC - Regional Commitee for Research Ethics)
Record Dates: First submitted 2016-07-29; First posted 2016-08-02 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Breast Cancer
Keywords: Telemark score, reliability
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- BCS: Photographs og consecutive group of 346 patients operated with breast conserving surgery were used to investigate cosmetic outcomes.
  Interventions: Other: digital photography
- DIEP: Photographs og consecutive group of 30 patients operated with DIEP-flap were used to assess cosmetic results
  Interventions: Other: digital photography

INTERVENTIONS:
Other: digital photography — Photographies with digital cameras were taken postoperatively for the documentation, anonymised and used for evaluation of cosmetic results after surgery.

SUMMARY:
This paper will present a specific tool for evaluation of cosmetic results after breast conserving surgery (BCS) and secondary breast reconstruction with free DIEP-flap. Introduction of a breast score system using digital photography seems to be a reliable tool for estimation of cosmetic results after breast surgery. The method has been employed on a specific group of 346 consecutive patients operated for breast cancer with breast conserving surgery. For the purpose of this study breast score system was tested on patients with free flap breast reconstruction (DIEP flap).

DETAILED DESCRIPTION:
Background: Validated instruments for assessing results after breast surgery are sparse. Investigators want to present a method used for the past 10 years at their institution for evaluation of the outcome after breast conserving surgery (BCS) and microsurgical breast reconstruction. Methods: 346 consecutive patients subjected to BCS for cancer and 30 patients operated with a deep inferior epigastric flap (DIEP ) were assessed at least one year after the operation. The Telemark Breast Score is a method based on standard two-dimensional photographs assessing the outcome after breast surgery in terms of volume, shape and symmetry. Three different panels including plastic surgeons, breast surgeons and nurses were invited to test the Telemark Breast Score. Consistency of agreement between and inside the panel groups was studied Results: Inter- and intra observer reliability was acceptable. Good stability of ratings could be shown in test-retests.

Conclusion: The Telemark Breast Scale is inexpensive, statistically reliable and can be applied for quality control after breast surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients operated for breast cancer at Hospital of Telemark

Exclusion Criteria:

* Patients operated for breast cancer and not subjected for irradiation

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 2 cohorts, one subjected to BCS and one to DIEP surgery.
Sampling Method: Non-Probability Sample
Enrollment: 376 (Actual)
Dates: Start 2014-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Telemark Breast Score | 2013-2014
  validation of Telemark Breast Score

IPD SHARING:
Plan to Share IPD: No